CLINICAL TRIAL: NCT00231907
Title: Influenza Vaccines: Mix and Match of Trivalent Inactivated Influenza (TIV) and Live Attenuated Influenza Vaccine (LAIV), a Phase I Safety, Immunogenicity, and Viral Shedding Study
Brief Title: A Phase I Safety and Immunogenicity Study of Mix and Match of Licensed Flu Vaccine and Flumist
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Robert Johnson, HHS/NIAID/DMID
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 04-101
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2010-08-27 (Estimated); Status verified 2010-02

CONDITIONS: Influenza
Keywords: influenza, vaccine, TIV, LAIV, booster, children
MeSH Terms: conditions — Influenza, Human | interventions — FluMist; Influenza Vaccines

ARMS (4):
- Vaccine 1: TIV. Vaccine 2: TIV. (Active Comparator): Vaccine 1: TIV. Vaccine 2: TIV.
  Interventions: Biological: Fluzone
- Vaccine 1: LAIV. Vaccine 2: TIV. (Experimental): Vaccine 1: LAIV. Vaccine 2: TIV.
  Interventions: Biological: FluMist; Biological: Fluzone
- Vaccine 1: LAIV. Vaccine 2: LAIV. (Experimental): Vaccine 1: LAIV. Vaccine 2: LAIV.
  Interventions: Biological: FluMist
- Vaccine 1: TIV. Vaccine 2: LAIV. (Experimental): Vaccine 1: TIV. Vaccine 2: LAIV.
  Interventions: Biological: FluMist; Biological: Fluzone

INTERVENTIONS:
Biological: FluMist — Live attenuated influenza vaccine (LAIV) containing approximately 10^7 TCID50 of each of the 3 influenza strains. 0.5 mL total dose volume administered intranasally via spray applicator (approximately 0.25 mL into each nostril). Administration of Flumist in children under 5 years of age is investigational.
  Arms: Vaccine 1: LAIV. Vaccine 2: LAIV.; Vaccine 1: LAIV. Vaccine 2: TIV.; Vaccine 1: TIV. Vaccine 2: LAIV.
Biological: Fluzone — Trivalent inactivated vaccine (TIV), licensed Fluzone preservative free pediatric dose, 0.25 mL administered intramuscularly to the anterolateral thigh muscle or deltoid muscle.
  Arms: Vaccine 1: LAIV. Vaccine 2: TIV.; Vaccine 1: TIV. Vaccine 2: LAIV.; Vaccine 1: TIV. Vaccine 2: TIV.

SUMMARY:
The purpose of this research is to compare the safety and ability to stimulate antibodies (part of the bodies proteins that fight infections) of two influenza (flu) vaccines given to children 12 to 35 months old. The two flu vaccines being compared are: trivalent inactivated influenza virus vaccine (TIV), a killed virus vaccine given as a shot licensed for use in children 6 months of age or older and live attenuated influenza vaccine (LAIV), a live (but weakened) virus vaccine licensed for children 5 years old and older given as a nose spray. The strains of the viruses have been weakened so that they do not cause typical influenza illness, but may allow the body to develop protection against the flu. LAIV vaccine is not licensed for children less than five years of age, therefore its use in this study is investigational. Participation is approximately 7 months in duration.

DETAILED DESCRIPTION:
This multi-site study is a phase I, open-label, 4-arm trial to evaluate 2 doses of influenza vaccine separated by 30 days. The vaccine will either be two doses of a single vaccine or a combination of vaccine products. FluMist®, a cold-adapted live attenuated influenza vaccine (LAIV), will be administered intranasally via spray applicator. Administration of FluMist in children less than 5 years of age is investigational. FluZone®, a trivalent inactivated influenza vaccine (TIV) licensed for use in children 6 months of age or older, will be administered intramuscularly (IM) to the anterolateral thigh muscle or deltoid muscle. Healthy children, ages 12 to 35 months old, who are representative of the population base of the vaccinating recruitment area, will be enrolled in this study at 3 sites. The primary study objective is to compare the safety and immunogenicity of two doses of licensed TIV or two doses of licensed LAIV with the safety and immunogenicity of a single dose of LAIV that is boosted with a dose of TIV versus children who receive an initial dose of TIV followed by a booster dose of LAIV among children 12 to 35 months of age. The secondary objective is to develop preliminary safety data on these combined vaccine regimes, and to evaluate the possibility that a single dose of TIV will either reduce the potential common side effects of LAIV or reduce the viral shedding associated with LAIV in children and to evaluate LAIV as a "primary" dose vaccine and TIV as a "booster vaccine" for inducing serum Hemagglutination Inhibition (HAI) antibodies. Vaccinees will be followed post-vaccination for safety, reactogenicity and immunogenicity. Patterns of viral shedding will be assessed 4 days after vaccination with LAIV. A final 6-month post-dose two vaccination contact will be made for serious adverse event data collection. Specifically, the investigators will assess the ability of LAIV to prime for a secondary immune response when TIV is given as a booster vaccine, and the investigators will evaluate TIV as a priming event for LAIV booster vaccine. Control groups will include TIV/TIV and LAIV/LAIV groups. The primary outcome measures for the study will be: assessment of post-dose 2 hemagglutination inhibition (HAI) antibodies to each of the 3 strains of influenza contained in the vaccine, safety assessment of each of the vaccines in combination vaccine. The secondary outcome measures include post-dose 1 HAI antibody titers and viral shedding after intranasal vaccination with live attenuated influenza vaccine. An additional secondary outcome will be assessment of secretory Immunoglobulin (Ig) A in nasal wash samples manifested after 1 or 2 doses of vaccine. An additional outcome will be Cell Mediated Immunity after 1 or 2 doses of vaccine. Blood will be collected on days 0, 30 and 60 for antibody detection. Nasal washes will be collected on day 0, 30 and 60 for secretory antibody measurements. A throat and nose swab sample will be collected on day 3 to 5 post LAIV vaccination to assess viral shedding and as dictated by presence of illness symptoms for viral culturing for two weeks after each dose of either LAIV or TIV vaccine. Up to 20 eligible participants will be enrolled in each of the 4 vaccination groups. As a four-arm trial with only active vaccine being administered by two different dosing routes, there will be no blinding to study assignment. Study duration is up to 3 years and individual participant duration is approximately 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Twelve to 35 months of age at enrollment.
* Minimum weight of 8 kg.
* In good health, as determined by parent/guardian verbal medical history and physical examination by clinical investigator.
* Parent/guardian available by telephone for safety data collection through 6 months post-dose 2.
* Ability of parent/guardian to understand and comply with the requirements of the protocol.
* Signed informed consent document and Health Insurance Portability and Accountability Act (HIPAA) authorization by the parent/guardian prior to performance of any study procedures.

Exclusion Criteria:

* History of hypersensitivity to any component of LAIV or TIV, including egg or egg products.
* History of hypersensitivity to gentamicin.
* Known or suspected immune deficiency diseases or immunosuppressed or have altered or compromised immune status as a consequence of treatment with immunosuppressive therapies.
* Known close contact with a severely immunocompromised person, such as someone currently in isolation secondary to a bone marrow transplantation (LAIV recipients should avoid close contact with severely immunocompromised individuals for at least 7 days after vaccination).
* History of chronic underlying medical conditions such as chronic disorders of the cardiovascular and pulmonary systems, chronic metabolic diseases (including diabetes), renal dysfunction, or hemoglobinopathies.
* History of Guillain-Barré syndrome.
* History of asthma or reactive airways disease.
* Acute febrile (>99.6 degrees Fahrenheit axillary) and/or respiratory illness, within the 72 hours prior to enrollment.
* Use of aspirin or aspirin containing products in the month prior to enrollment or anticipated use during the study.
* Administration of any intranasal medication within 2 weeks prior to enrollment or expected receipt during this study.
* Previous receipt of an influenza vaccine.
* Administration of any live virus vaccine within 4 weeks prior to enrollment or (other than study vaccine) planned receipt of another live virus vaccine before completion of the 2 weeks after the last vaccination in this study*
* Administration of any inactivated vaccine within 2 weeks prior to enrollment or planned receipt of another inactivated vaccine before 2 weeks after the last vaccination in this study*
* Participation in another investigational trial or administration of any investigational drug within 1 month prior to enrollment or during this study.
* Any condition that in the opinion of the investigator would interfere with the interpretation or evaluation of the vaccine.

  * Routine immunizations can be resumed after the memory aid period following dose 2.

Ages: 12 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2005-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Assessment of post-dose 2 HAI (Hemagglutination Inhibition) antibodies to each of the 3 strains of influenza contained in the vaccine. | Blood sample taken on day 0, 28 + 7, day 60 +/- 4.
Safety assessment of each of the vaccines in combination vaccine. | Duration of study.

SECONDARY OUTCOMES:
Assessment of secretory IgA in nasal wash samples manifested after 1 or 2 doses of vaccine. | Nasal wash samples will be colllected on Days 0, 30, and 60.
CMI | Blood sample taken on Day 0, Day 28 + 7, Day 60 +/- 4.
Post-dose 1 HAI (Hemagglutination Inhibition) antibody titers and viral shedding. | Day 3 to 5 post LAIV vaccination.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Saint Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Derived] Hoft DF, Babusis E, Worku S, Spencer CT, Lottenbach K, Truscott SM, Abate G, Sakala IG, Edwards KM, Creech CB, Gerber MA, Bernstein DI, Newman F, Graham I, Anderson EL, Belshe RB. Live and inactivated influenza vaccines induce similar humoral responses, but only live vaccines induce diverse T-cell responses in young children. J Infect Dis. 2011 Sep 15;204(6):845-53. doi: 10.1093/infdis/jir436. Epub 2011 Aug 15. PMID 21846636